CLINICAL TRIAL: NCT05259553
Title: Evaluation of Predictive Biomarkers in de Novo Multiple Myeloma on the Onset of Venous Thromboembolism, Its Impact on Clinical Outcome and Thromboprophylaxis (VESICOM)
Brief Title: Biomarkers in Multiple Myeloma
Acronym: VESICOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-0701; 2021-A01895-36 (Other: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hematological Patients; Newly Diagnosed Multiple Myeloma; Chemotherapy
Keywords: hematology; multiple myeloma; chemotherapy; thromboprophylaxis
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with multiple myeloma (Experimental): Adult patient, over 18 years old, with newly diagnosed multiple myeloma, indication of chemotherapy.
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Peripheral blood sampling will be performed at different time points of the study, for a total volume of 20-40 mL:
  * Sampling before MM treatment,
  * Sampling during MM treatment (at 3 months post-initiation if no autograft or before autograft),
  * Only for Patients treated with Apixaban or Eliquis®, 2 additional samplings during MM treatment for pharmacokinetics analysis.

SUMMARY:
The association between multiple myeloma (MM) and venous thromboembolism (VTE) is well known. Indeed, the incidence of VTE is increased in patients with newly diagnosed MM and in patients treated by immunomodulatory drugs in combination with glucocorticoids. Moreover, the clinical outcome of MM is supposed to be correlated to the risk of thrombosis. At the biological level, a number of hemostasis abnormalities participate in increasing VTE incidence. Yet, data on predictive biomarkers linked to VTE are limited.

DETAILED DESCRIPTION:
There is a need to discern predictive biomarkers in order to better identify patients at risk of developing VTE, to decipher the mechanisms by which myeloma treatments interfere and in fine to choose an adequate thromboprophylaxis. In this context, it is important to document the precise expression of coagulation factors and to profile point-of-care tests for coagulation monitoring in newly diagnosed MM patients, before and during treatment. In addition, thromboprophylaxis is systematically included in therapeutic MM strategies, especially direct oral anticoagulants, without knowing whether potential drug interactions are occurring. This study aims at evaluating and validating predictive biomarkers of VTE in MM, and at identifying patients whose thromboprophylaxis is required and may potentially be adjusted because of drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to a social security regimen or beneficiary of the same
* Signed written informed consent form
* Confirmed diagnosis of de novo multiple myeloma, non-previously treated and requiring treatment.

Exclusion Criteria:

* Pregnant women
* Patient under guardianship or deprived of his liberty or any condition that may affect the patient's ability to understand and sign the informed consent
* Refusing participation
* Patient whose follow-up or life expectancy is less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Level of thrombin generation in newly diagnosed and untreated MM | 24 months
  Measurement of thrombin on plasma from newly diagnosed MM patients before the initiation of chemotherapy
Level of factor VIII in newly diagnosed and untreated MM | 24 months
  Measurement of factor VIII on plasma from newly diagnosed MM patients before the initiation of chemotherapy
Level of D-Dimers in newly diagnosed and untreated MM | 24 months
  Measurement of D-Dimers on plasma from newly diagnosed MM patients before the initiation of chemotherapy
Level of pro-coagulant phospholipids in newly diagnosed and untreated MM | 24 months
  Measurement of pro-coagulant phospholipids on plasma from newly diagnosed MM patients before the initiation of chemotherapy

SECONDARY OUTCOMES:
Association between biomarkers (thrombin, factor VIII, D-Dimers, pro-coagulant phospholipids) and VTE onset | 24 months
  Correlation between the plasma level of biomarkers and clinical data
Association between biomarkers (thrombin, factor VIII, D-Dimers, pro-coagulant phospholipids) and MM outcome | 24 months
  Correlation between the plasma level of biomarkers and clinical data
Evolution of biomarkers (thrombin, factor VIII, D-Dimers, pro-coagulant phospholipids) at 3 months post-treatment | 24 months
  Correlation between the plasma level of biomarkers and clinical data
Evaluation of the exposition of Apixaban (Eliquis®) | 24 months
  Plasma level of Apixaban in MM treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Chalayer, MD, Principal Investigator — CHU de Saint-Etienne
Locations (2):
- France (2):
  - Hospices Civils de Lyon, Lyon
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No